CLINICAL TRIAL: NCT06371274
Title: Efficacy and Safety Study of Oral All-trans Retinoic Acid Combined With Toripalimab in Patients With Inoperable Locally Advanced, Recurrent, or Metastatic Triple-negative Breast Cancer Who Had Failed Prior Second-line or Higher Standard Therapy.
Brief Title: A Study on the Efficacy and Safety of Oral All-trans Retinoic Acid Combined With Toripalimab in TNBC.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Shanghai Longfine Biotechnology Co., Ltd. (Unknown); TopAlliance (Unknown)
Responsible Party: Principal Investigator, Jian Liu, chief pharmacist, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZYYY-IIT-TNBC-001
Record Dates: First submitted 2024-04-02; First posted 2024-04-17 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Triple-negative Breast Cancer
Keywords: all-trans retinoic acid; Toripalimab; triple-negative breast cancer; efficacy; safety
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ATRA+Toripalimab (Experimental): Eligible participants are subjected to take all-trans retinoic acid orally at a dose of 150 mg/m2 per day, twice a day for three consecutive days per cycle (d0~d2), and intravenous infusion of PD-1 monoclonal antibody at a dose of 240 mg on day 1 of each cycle (d1), with cycles repeated every 3 weeks until disease progression, death, loss to follow-up, intolerable toxicity, or meeting other withdrawal or termination criteria (whichever occurs first), for a maximum duration of 2 years.
  Interventions: Drug: ATRA; Drug: Toripalimab

INTERVENTIONS:
Drug: ATRA — ATRA is the main active metabolite of vitamin A. Studies have shown that ATRA can also reduce the number of MDSC in solid tumor patients, promote their differentiation and maturation, remove the immunosuppressive ability of MDSC, improve the tumor immune microenvironment, and thus improve the tumor treatment efficacy.
Drug: Toripalimab — Toripalimab is a fully human monoclonal antibody injection against PD-1 receptor. The NMPA has accepted the application of Toripalimab for a new indication for the treatment of initial metastatic or relapsed metastatic TNBC with PD-L1 positive (CPS≥1).

SUMMARY:
To evaluate the clinical efficacy and safety of oral all-trans retinoic acid in combination with toripalimab in patients with locally advanced, recurrent, or metastatic triple-negative breast cancer who had failed second-line and subsequent therapy.

DETAILED DESCRIPTION:
The study is designed as a single arm, open-label, mono-center exploratory trial, aiming to evaluate the clinical efficacy and safety of oral all-trans retinoic acid in combination with toripalimab in patients with locally advanced, unresectable, recurrent, or metastatic triple-negative breast cancer who had failed second-line and subsequent standard treatments. 32 subjects are planned to be enrolled. Eligible participants are subjected to take all-trans retinoic acid orally at a dose of 150 mg/m2 per day, twice a day for three consecutive days per cycle (d0~d2), and intravenous infusion of PD-1 monoclonal antibody at a dose of 240 mg on day 1 of each cycle (d1), with cycles repeated every 3 weeks until disease progression, death, loss to follow-up, intolerable toxicity, or meeting other withdrawal or termination criteria (whichever occurs first), for a maximum duration of 2 years. Each subject's study process includes a screening period (within 28 days), a treatment period, and a follow-up period. Subjects will sign the informed consent form and complete all baseline assessments during the screening period. Qualified subjects will enter the treatment period, followed by the survival follow-up every 3 months after the completion of the treatment period. Tumor assessments (contrast-enhanced CT) will be conducted every 2 cycles (6 weeks) during the combination treatment period, and efficacy evaluation will be based on RECIST 1.1 criteria. Moreover, iORR and iPFS were assessed by investigators based on iRECIST criteria. Adverse events will be assessed using NCI-CTCAE version 5.0, with observation of adverse events up to 30 days after the last treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of signing the informed consent form;
2. Pathologically confirmed as triple-negative breast cancer based on recent biopsy or other pathological specimens, with histological and/or cytological diagnosis;
3. Patients with unresectable locally advanced or metastatic triple-negative breast cancer who have failed at least second-line standard treatment regimens;
4. According to RECIST 1.1, at least one measurable lesion is required. Patients with only skin lesions or bone lesions are not eligible for inclusion;
5. Adequate organ and bone marrow function (not received blood transfusions, recombinant human platelet growth factor, or colony-stimulating factor treatment in the 2 weeks before screening);
6. The subject voluntarily agrees to participate in this study, signs the informed consent form, and is able to comply with the visits and related procedures specified in the protocol.

Exclusion Criteria:

1. Known symptomatic or uncontrolled brain metastasis or other central nervous system (CNS) metastases;
2. Patients with other malignant tumors, excluding those with cured basal cell or squamous cell skin carcinoma or in situ cervical cancer. Patients with other malignant tumors must have a disease-free interval of at least 5 years;
3. Any severe and/or uncontrolled concurrent illness that hinders the patient's participation in the study;
4. History of immunodeficiency, autoimmune diseases, the need for immunosuppressive therapy (daily dose >10 mg of prednisone or equivalent), or a history of chronic infections;
5. History of deep vein thrombosis or pulmonary embolism;
6. Severe osteoporosis or patients with bone metastases;
7. Participants who, within the first 4 weeks before the initiation of the study treatment or during the 5 half-lives of any drugs used in the pre-study period (whichever is shorter), have received any chemotherapy, immunotherapy, biologic therapy, or participated in other drug clinical trials, or received traditional Chinese medicine preparations for the treatment of approved anticancer indications or radiotherapy within the first 2 weeks before the initiation of the study treatment, or have undergone major surgery within the first 4 weeks before the initiation of the study treatment;
8. Patients with active hepatitis B or C; known history of human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS); positive syphilis antibody test;
9. History of severe drug allergies or known allergy to any component of the investigational drug as per the prescription;
10. The investigator considers the participant unsuitable for the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 29 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 2 years
  During the combined therapy, tumor assessment (enhanced CT) is conducted every 2 cycles (6 weeks), and the efficacy is evaluated using the RECIST 1.1 criteria. ORR will be summarized as the proportion of subjects achieving objective tumor responses (complete response or partial response). ORR and its 95% confidence interval will be calculated.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | up to 2 years
  PFS defined as the time from enrollment until disease progression or death (whichever occurs first).
Duration of Response (DOR) | up to 2 years
  For responders (complete response or partial response), DOR is defined as the time from the earliest date meeting the response criteria to disease progression or death for any reason (whichever occurs first). For subjects who do not experience progression after meeting response criteria and continue to survive, DOR will be censored at the last evaluable tumor assessment date or the last follow-up date for disease progression.
Overall Survival (OS) | up to 2 years
  OS is defined as the time interval between the date of the first dose and the date of death for any reason. Kaplan-Meier methodology will be used to estimate median OS, OS rates, and their 95% confidence intervals at different time points.

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse events as assessed by NCI-CTCAE 5.0 | up to 2 years
  Adverse events and toxicity will be assessed according to the NCI-CTCAE 5.0 criteria. Medical review of adverse events and laboratory values will be conducted, and a safety assessment will be completed. Adverse events occurring after treatment will be summarized based on preferred terms, organ system classification, NCI-CTCAE severity grading, and their relationship to the investigational therapy. Safety assessments will be conducted for all subjects receiving the study drug, with evaluation starting from the date of informed consent signing and continuing until the study concludes or 30 days after drug discontinuation.
Exploratory biomarkers-peripheral blood lymphocyte analysis | start from the time of enrollment to the end of the study, assessed up to 2 years
  Whole blood samples will be collected during the cycle 1 treatment period, defined as before the ATRA first dose (d0), d1, d2, d7 and d14. Later, the biological sample will also be provided before following each cycle treatment as only the subjects who have given informed consent and are willing to provide. Peripheral blood mononuclear cells (PBMCs) will be isolated and subjected to flow cytometry analysis using myeloid-derived suppressor cell (MDSC) and T lymphocyte molecular markers. Changes in the quantity, subsets, and surface markers of MDSC before and after treatment will be evaluated, and their relationship with the combined treatment response will be assessed.
Exploratory biomarkers-Serum Metabolomics Analysis | start from the time of enrollment to the end of the study, assessed up to 2 years
  Plasma samples will be collected during the cycle 1 treatment period, defined as before the ATRA first dose (d0), d1, d2, d7 and d14. Later, the biological sample will also be provided before following each cycle treatment as only the subjects who have given informed consent and are willing to provide. The Q300 metabolomics chip will be employed to quantitatively measure the concentrations of various metabolites. Data analysis will utilize correlation analysis methods (Pearson correlation) to assess the correlation between changes in metabolites and immune cell activity, as well as potential clinical efficacy, aiming to explore potential biomarkers for the combined treatment.
Exploratory biomarkers-Fecal Microbiota Analysis | start from the time of enrollment to the end of the study, assessed up to 2 years
  Fecal samples will be collected during the cycle 1 treatment period, defined as before the ATRA first dose (d0), d1, d7 and d14. Later, the biological sample will also be provided before following each cycle treatment as only the subjects who have given informed consent and are willing to provide. Classification and identification of the intestinal microbiota will be performed. Depending on the data type, chi-square tests, t-tests, or other non-parametric tests will be selected to compare differences between groups with different efficacy responses.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaochen Zhang, MD, Principal Investigator — Zhejiang University
Locations (1):
- The first affiliated hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang Province, P.R. China, China

IPD SHARING:
Plan to Share IPD: No